CLINICAL TRIAL: NCT06468033
Title: A Randomized, Double-Blind, Placebo-Controlled Multicenter Phase III Study to Assess Efficacy and Safety of Ropeginterferon Alfa-2b (P1101) in Adult Patients With Pre-fibrotic/Early Primary Myelofibrosis (PMF) or Overt PMF at Low or Intermediate-1 Risk According to DIPSS Plus (HOPE-PMF): The Core Study and Its Extension Study
Brief Title: P1101 in Treating Patients With Early PMF or Overt PMF at Low or Intermediate-1 Risk
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: PharmaEssentia (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: A23-302
Record Dates: First submitted 2024-06-10; First posted 2024-06-21 (Actual); Last update posted 2025-08-13 (Actual); Status verified 2025-08

CONDITIONS: Primary Myelofibrosis; Myeloproliferative Neoplasm
Keywords: P1101; Primary Myelofibrosis; PMF; Ropeginterferon; PharmaEssentia; Myeloproliferative neoplasms; MPN; Pre-fibrotic; Low or Intermediate-1 Risk
MeSH Terms: conditions — Primary Myelofibrosis; Myeloproliferative Disorders

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Double-Blind
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Ropeginterferon alfa-2b (P1101) (Experimental): Ropeginterferon alfa-2b (P1101) is administrated subcutaneously (SC) every two weeks (± 3 days) until 80 weeks.
  Interventions: Biological: Ropeginterferon alfa-2b
- Placebo control (Placebo Comparator): Placebo is administrated subcutaneously (SC) every two weeks (± 3 days) until 80 weeks.
  Interventions: Other: Placebo

INTERVENTIONS:
Biological: Ropeginterferon alfa-2b — Pre-filled Syringe.
  Dosage: up to 500mcg
  Other Names: P1101
  Arms: Ropeginterferon alfa-2b (P1101)
Other: Placebo — Placebo is a look-alike substance with the intervention (Ropeginterferon alfa-2b) that contains no active drug.
  Arms: Placebo control

SUMMARY:
This is a phase 3 double-blind clinical trial arm to test Ropeginterferon alfa-2b (P1101) in adult patients with Primary Myelofibrosis (PMF) at early stage or low to medium risk.

Participants will receive the study drug/placebo bi-weekly and have an assessment visit every 4 weeks. The ratio of study drug to placebo group is 2:1.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female patients aged ≥18 years at the time of signing the informed consent form;
2. Patients with pre-fibrotic/early PMF (Pre-PMF) or overt primary myelofibrosis at low to intermediate-1 risk according to DIPSS plus, diagnosed according to WHO 2016 or 2022 classification;
3. With good liver function at screening, which is defined as total bilirubin ≤1.5 × upper limit of normal (ULN), international normalized ratio (INR) ≤1.5 × ULN, albumin >3.5 g/dL, alanine aminotransferase (ALT) ≤2.0 × ULN, and aspartate aminotransferase (AST) ≤2.0 × ULN;
4. Hgb ≥10.0 g/dL at screening;
5. Neutrophil count ≥1.0 × 10^9/L at screening;
6. Creatinine clearance rate ≥30 mL/min at screening (according to the Cockcroft-Gault formula);
7. Females of childbearing potential, as well as all women <2 years after the onset of menopause, must agree to use an acceptable form of birth control until 60 days following the last dose of the study drug, and females must agree to not breastfeed during the study;
8. Written informed consent obtained from the subject and ability for the subject to comply with the requirements of the study.

Exclusion Criteria:

1. Any known contraindications to interferon α or hypersensitivity to interferon α;
2. Patients with prior interferon therapy having poor tolerability or lack of efficacy to the previous interferon therapy per investigator's judgement;
3. Patients with an ongoing cytoreduction (e.g., HU or IFN-α) at the time of screening if, in the Investigator's opinion, randomizing them into the placebo arm will lead to immediate rebound increase of peripheral blood counts and thus may jeopardize their health status;
4. With severe or serious diseases that, in the Investigator's opinion, may affect the patient's participation in this study;
5. History of major organ transplantation;
6. Pregnant or breastfeeding women;
7. Patients with any other diseases that will affect the study results or may weaken the compliance to protocol per the Investigator's judgment;
8. Use any investigational drug <4 weeks prior to the first dose of study drug, or not recovered from effects of prior administration of any investigational drug.
9. Eligible for JAK inhibitor therapy at screening.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 150 (Estimated)
Dates: Start 2025-07-18 (Actual); Primary Completion 2027-09-30 (Estimated); Study Completion 2028-09-30 (Estimated)

PRIMARY OUTCOMES:
Number of Participants with Platelet count equal or less (≤) 400 × 10^9/L | 80 weeks
  Platelet count ≤400 × 10^9/L is one of the criteria for clinically relevant complete hematologic response (CrCHR).
Number of Participants with White Blood Cells (WBC) count equal or less (≤) 10 × 10^9/L | 80 weeks
  White Blood Cells (WBC) count ≤10 × 10^9/L is one of the criteria for clinically relevant complete hematologic response (CrCHR).
Number of Participants with Hemoglobin (Hgb) equal or greater (≧) 10.0 g/dL | 80 weeks
  Peripheral blood: Hemoglobin (Hgb) ≧ 10.0 g/dL is one of the criteria for clinically relevant complete hematologic response (CrCHR).
Number of Participants absence of major thrombotic events | 80 weeks
  The absence of major thrombotic events during the observation time frame is one of the criteria for clinically relevant complete hematologic response (CrCHR).
Number of Participants with no progression to secondary acute myeloid leukemia (AML). | 80 weeks
  The absence of progression to secondary acute myeloid leukemia (AML) is one of the criteria for clinically relevant complete hematologic remission (CrCHR).
Number of Participants with no progression on the Total Symptom Score (TSS) | 80 weeks
  The TSS score is utilized to evaluate clinical symptoms, which is based on the MFSAF Total Symptom Score (TSS) form v4.0.
  No progression is defined as:
  * The participants who still have a TSS score equal to or less than (≤) 10 If the baseline score is ≤ 10.
  * The participants with a TSS score no increase than 50% If the baseline score is greater than (>) 10.

CONTACTS AND LOCATIONS:
Overall Officials: Toshiaki Sato, MD/PhD, Study Director — PharmaEssentia JP
Locations (1):
- University of Yamanashi Hospital, Chūō, Yamanashi, Japan